CLINICAL TRIAL: NCT00329277
Title: Detection of Topographic Residual Acuity in Patients With Age Related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNM200601
Record Dates: First submitted 2006-05-23; First posted 2006-05-24 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2006-11

CONDITIONS: Age-Related Macular Degeneration
Keywords: age-related macular degeneration; preferred retinal locus; macular perimetry
MeSH Terms: conditions — Macular Degeneration

INTERVENTIONS:
Procedure: perimetry

SUMMARY:
Standard perimetry provides information on topographical retinal sensitivity to light stimuli, however the said locus is not necessarily the preferred locus for fixation. Standard perimetry could also be used as a way for macular scotoma mapping, indirectly showing the fixation locus. Topographic acuity at the preferred retinal locus can be determined if correlation between loci with high sensitivity, eccentric fixation loci and potential visual acuity measurements are correlated.

PURPOSE OF THE STUDY:

Determination of visual acuity at preferred retinal locus in Low Vision patients with ARMD using eye standard automated and computerized perimetry methods.

ELIGIBILITY:
Inclusion Criteria:

* AMD with documented pathology
* Low Vision both eyes
* BCVA 20/50-20/400 in best eye

Exclusion Criteria:

* Cognitive impairment
* Other retinal pathology
* Previous retinal surgery
* Significant media opacity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Location of eccentric retinal locus of highest fixation accuracy

SECONDARY OUTCOMES:
Location of eccentric locus with best retinal sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Markowitz, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Dr S N Markowitz, Toronto, Ontario, Canada